CLINICAL TRIAL: NCT06977828
Title: A Prospective, Single-arm, Phase II Clinical Study of Tislelizumab Combined With Anlotinib and Platinum-based Doublet Perioperative Therapy for Resectable Stage II-IIIB Driver Gene-negative NSCLC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Lingxiang Liu, MD, The First Affiliated Hospital with Nanjing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-SR-259
Record Dates: First submitted 2025-05-11; First posted 2025-05-18 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: NSCLC (Non-small Cell Lung Cancer); Neoadjuvant Immunotherapy; Adjuvant Immunotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — tislelizumab; anlotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- tislelizumab in combination with anlotinib and platinum-based doublet chemotherapy (Experimental)
  Interventions: Drug: tislelizumab in combination with anlotinib and platinum-based doublet chemotherapy

INTERVENTIONS:
Drug: tislelizumab in combination with anlotinib and platinum-based doublet chemotherapy — After receiving 4 cycles of tislelizumab combined with anlotinib and platinum-based doublet chemotherapy, the subjects will be evaluated by a multidisciplinary team (MDT) to determine whether to proceed with radical surgical resection. The surgery will be performed within 3 to 7 weeks after the last neoadjuvant treatment. Postoperatively, patients will be divided into two subgroups based on the pathological results: For patients with postoperative pathological pCR, tislelizumab monotherapy will be used for maintenance treatment; For patients with postoperative pathological non-pCR, tislelizumab combined with anlotinib will be used for maintenance treatment. Both groups will continue treatment until disease progression, intolerable toxicity, withdrawal of informed consent, initiation of other anti-tumor therapy, death, or other situations specified in the protocol that require treatment cessation, whichever occurs first. The maximum treatment duration is 12 months

SUMMARY:
The goal of this clinical trial is to learn if tislelizumab in combination with anlotinib and platinum-based doublet chemotherapy works to treat for resectable stage II-IIIB driver gene-negative NSCLC. It will also learn about the safety of tislelizumab in combination with anlotinib and platinum-based doublet chemotherapy.

The main questions it aims to answer are:

1. Does tislelizumab combined with anlotinib and platinum-based doublet perioperative therapy can increase pCR rate as well as MPR rate、EFS、DFS、ORR、OS for resectable stage II-IIIB driver gene-negative NSCLC?
2. Is tislelizumab combined with anlotinib and platinum-based doublet perioperative therapy safe?

Participants with histologically or cytologically confirmed NSCLC, potentially resectable, driver gene negative (II- IIIB stage), and without prior systemic treatment, who have signed the informed consent, will be screened for inclusion. After receiving 4 cycles of tislelizumab combined with anlotinib and platinum-based doublet chemotherapy, the subjects will be evaluated by a multidisciplinary team (MDT) to determine whether to proceed with radical surgical resection. The surgery will be performed within 3 to 7 weeks after the last neoadjuvant treatment. Postoperatively, patients will be divided into two subgroups based on the pathological results: For patients with postoperative pathological pCR, tislelizumab monotherapy will be used for maintenance treatment; For patients with postoperative pathological non-pCR, tislelizumab combined with anlotinib will be used for maintenance treatment. Both groups will continue treatment until disease progression as defined by RECIST 1.1, intolerable toxicity, withdrawal of informed consent, initiation of other anti-tumor therapy, death, or other situations specified in the protocol that require treatment cessation, whichever occurs first. The maximum treatment duration is 12 months. Survival and safety assessments will be continuously conducted thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Fully understand and voluntarily sign the informed consent for this study;
* Age ≥18 years old and ≤75 years old, male or female;
* Patients with histologically or cytologically confirmed resectable stage II-IIIB non-small cell lung cancer;
* ECOG 0-1;
* No EGFR sensitive mutation, ALK or ROS1 fusion mutation was confirmed by tissue genetic testing before enrollment.
* Had not received any previous systemic treatment for non-small cell lung cancer;
* Patients with normal organ function within 7 days before enrollment met the following criteria:

  1. Blood routine test (no blood transfusion history within 14 days) :
  2. Hemoglobin (HB)≥90g/L; Absolute neutrophil count (ANC)≥1.5×109/L; j Platelet count (PLT)≥80×109/L.
  3. Biochemical test results met the following criteria:

     Total bilirubin (TBIL)≤1.5 ULN; Alanine aminotransferase (ALT) and aspartate aminotransferase (AST)≤2.5 ULN, or 5 ULN if liver metastasis occurs; Serum creatinine (Cr)≤1.5 ULN or creatinine clearance (CCr)≥60mL/min. Left ventricular ejection fraction (LVEF)≥50%; Urine routine examination showed urine protein < 2+ or 24-hour urine protein < 1g; Serum amylase and lipase ≤ ULN.
* Male or female patients of childbearing potential voluntarily use an effective method of contraception, such as dual barrier methods, condoms, oral or injectable contraceptives, intrauterine devices, etc. during the study and for 6 months after the last study medication. All female patients will be considered fertile unless they have undergone natural menopause, artificial menopause, or sterilization (e.g., hysterectomy, bilateral adnophorectomy, or radioactive ovarian irradiation).

Exclusion Criteria:

* The pathological types of the patients were mixed with components of small cell lung cancer, neuroendocrine carcinoma, sarcoma, salivary gland tumor and mesenchymal tumor.
* Central, caenorrhea squamous cell carcinoma or hemoptysis non-small cell lung cancer (hemoptysis >50 mL/ day);
* The tumor is surrounded by large blood vessels, and there is a potential risk of hemoptysis after anlotinib treatment;
* Presence of symptomatic or clinically significant thyroid dysfunction at screening (hypothyroidism controlled only with thyroid hormone replacement could be included);
* Patients who have been diagnosed with immunodeficiency or are receiving systemic glucocorticoid therapy or any other form of immunosuppressive therapy (prednisone at a dose of >10mg/ day or other equivalent efficacy hormone) and continue to use it within 2 weeks before the first dose;
* Active autoimmune disease requiring systemic therapy (e.g., disease-modifying medications, corticosteroids, or immunosuppressive agents), including but not limited to inflammatory bowel disease such as ulcerative colitis or Crohn's disease, occurred within 2 years before enrollment; Diverticulitis; Celiac disease; Systemic lupus erythematosus; Sarcoidosis syndrome or Wegener syndrome (granulomatosis with polyangiitis); Graves' disease; Rheumatoid arthritis; Multiple sclerosis; Vasculitis; Glomerulonephritis; Antiphospholipid syndrome; Hypophysitis; Uveitis and so on. Alternative therapies (e.g., thyroxine, insulin, or physiological doses of corticosteroids for adrenal or pituitary insufficiency) were not considered systemic treatments. Patients who were positive for autoimmune antibodies were eligible for enrollment after investigator evaluation to confirm the absence of autoimmune disease requiring systemic treatment. ;
* Vaccination or attenuated vaccine within 4 weeks before enrollment;
* Received approved or investigational systemic anti-tumor therapy within 4 weeks before enrollment, including chemotherapy, radical radiotherapy, biological immunotherapy, targeted therapy, and traditional Chinese medicine therapy (traditional Chinese medicine therapy with clear indications for anti-tumor, after a 3-week washout period can also be enrolled);
* Participated in clinical trials of other drugs not yet approved or marketed in China and received treatment with corresponding drugs within 4 weeks before enrollment;
* Patients who underwent major surgery or unhealed wounds, ulcers, or fractures within 4 weeks before enrollment;
* International normalized ratio (INR) >1.5 or activated partial prothrombin time (APTT) >1.5×ULN; twelve Electrolyte abnormalities that were judged by the investigator to be clinically significant;
* Patients have drug-uncontrolled hypertension defined as systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg;
* The patient has any current disease or condition that affects drug absorption or the patient is unable to take anlotinib orally;
* Patients with active gastric and duodenal ulcer, ulcerative colitis and other gastrointestinal diseases or unresected tumors with active bleeding, or other conditions that may cause gastrointestinal bleeding or perforation as judged by the investigators;
* Patients with evidence or history of significant bleeding tendency within 3 months before enrollment (bleeding >30 mL within 3 months, hematemesis, melena, hematochezia), hemoptysis (>5 mL of fresh blood within 4 weeks) or thromboembolic events (including stroke events and/or transient ischemic attack) within 12 months;
* Grade 1 or above myocardial ischemia, myocardial infarction or severe arrhythmia (including QTc≥450 ms(male), QTc≥ 470ms(female) and NYHA class 1 or above congestive heart failure;
* Other malignant tumors in the past 5 years, excluding basal cell or squamous cell carcinoma of the skin after radical resection, or carcinoma in situ of the cervix;
* Severe active or uncontrolled infection (≥CTCAE v5.0 grade 2 infection);
* Known human immunodeficiency virus (HIV) infection; A known history of clinically significant liver disease, including viral hepatitis (known hepatitis B virus (HBV) carriers must rule out active HBV infection, defined as HBV DNA positivity (>1×104 copies /mL or >2000 IU/ml); Known hepatitis C virus (HCV) infection and HCV RNA positive (>1×103 copies /mL), or other hepatitis, liver cirrhosis] (excluding patients with previous antiviral treatment, the relevant test results returned to normal);
* Tuberculosis that is active or currently in need of medical intervention, including but not limited to tuberculosis;
* A history of acute or chronic pancreatitis, pancreatic surgery, or risk factors that may increase the risk of pancreatitis;
* Has not fully recovered from any intervention-induced toxicity and/or complications before enrollment (i.e., > grade 1 or not recovered to baseline required levels);
* Women who are pregnant (positive pregnancy test before medication) or breastfeeding;
* Received blood transfusion, blood products, and hematopoietic factors such as albumin and granulocyte colony-stimulating factor (G-CSF) within 14 days before enrollment;
* Brachytherapy (radioactive seed implantation) within 60 days before enrollment;
* Known response to tislelizumab and/or chemotherapy of choice (non-squamous NSCLC: pemetrexed plus cisplatin or carboplatin; Squamous NSCLC: allergic reaction to the active ingredient and/or any excipients of paclitaxel or albumin paclitaxel plus cisplatin or carboplatin);
* Any other medical condition, clinically significant metabolic, physical or laboratory abnormality, medical history, disease, treatment or laboratory abnormality that may interfere with the results of the trial or prevent the subject from participating fully in the study, in the investigator's judgment, There is a reason to suspect that the patient has a disease or condition (e.g., having seizures and requiring treatment) that would be inappropriate for the study drug, that would affect the interpretation of the study results, or that the investigator believes that participation in the study would not be in the subject's best interest;
* The presence of any clinically significant systemic disease that is judged by the investigator to require treatment, including but not limited to thyroid disease (patients with stable thyroid function after hormone replacement therapy can be enrolled), organ transplant recipient, history of mental illness, and history of drug abuse/addiction, alcohol or drug abuse;
* Local or systemic disease that is not caused by malignancy, or a secondary reaction to cancer, and may result in a high medical risk and/or uncertainty in the evaluation of survival.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07-20 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Pathological Complete Response (pCR) rate | Up to ~64 months
  Pathological complete response (pCR) is measured as the percentage of participants with a pathological complete response as assessed by the central pathologist at the time of definitive surgery. pCR is defined as having no residual invasive squamous cell carcinoma within the resected primary tumor specimen and all sampled regional lymph nodes.

SECONDARY OUTCOMES:
Major Pathological Response (mPR) rate | Up to ~64 months
  The percentage of participants with a major pathological response (mPR) as assessed by the Central Pathologist at the time of definitive surgery. mPR is defined as ≤10% invasive squamous cell carcinoma within the resected primary tumor specimen and all the sampled regional lymph nodes.
Event-free Survival (EFS) | Up to ~80 months
  EFS is the time from the date of randomization to the date of first record of any of the following events: radiographic disease progression; local or distant progression or recurrence as assessed with imaging or biopsy as indicated; or death due to any cause. Radiographic disease progression during neoadjuvant phase that precludes surgery will be considered an event; a secondary malignancy will not be considered an event.
Disease-free survival (DFS) | Up to ~80 months
  defined as the period from the first day after radical surgery (when the disease is confirmed to be cured) to local recurrence or distant metastasis or the time of death for any reason was determined by the investigator during the period of adjuvant therapy and safety follow-up, whichever occurred first.Only patients who underwent R0 resection will be analyzed.
Objective response rate (ORR) | Up to ~64 months
  defined as the proportion of all patients with measurable disease at baseline as assessed by the investigator according to RECIST version 1.1 who achieved a complete response (CR) or partial response (PR). The proportion of patients achieving complete remission (CR) or partial remission (PR) among the patients
Overall survival (OS) | Up to ~92 months
  It is defined as the time from the date of patient enrollment to the date of death due to any cause.
Percentage of Participants Experiencing An Adverse Event (AEs) | From time of first dose of study treatment until the end of follow-up (up to ~92 months)
  Percentage of participants experiencing any sign, symptom, disease, or worsening of preexisting condition temporally associated with study therapy and irrespective of causality to study therapy

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No